CLINICAL TRIAL: NCT01186016
Title: Developing Genetic Education for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0226-09-FB; 1R21DK084517-01 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-08-20 (Estimated); Results first posted 2022-12-07 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Smoking
Keywords: Genetic Education; Smoking Cessation; Quitting Smoking; Standard Smoking Cessation Program; Genetic Education for Smoking Cessation
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic Education Session (GES) (Experimental): The objectives are to: discuss the impact of the human genome project; define basic genetic concepts and terminology; distinguish between single-gene and multifactorial genetic diseases/conditions; describe genetic counseling/testing; identify uses of pharmacogenetics; discuss psychological and legal/ethical implications of genetic discoveries; smoking as a multifactorial behavior; findings of epidemiological studies about smoking heritability; research about candidate genotypes DRD2 and CYP2A6; and potential use of genotyping to tailor smoking cessation treatment. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of OTC transdermal nicotine replacement therapy.
  Interventions: Behavioral: Genetic Education Session
- Nutrition Education Session (NES) (Active Comparator): The objective is to provide a control group that will received comparable attention as the experimental group by providing USDA approved nutritional information (MyPyramid) dietary and food safety guidelines. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of OTC transdermal nicotine replacement therapy.
  Interventions: Behavioral: Nutrition Education Session

INTERVENTIONS:
Behavioral: Genetic Education Session — The intervention includes receiving education about genetics and smoking. The content is basic genetics and education about the multifactorial nature of smoking; research findings about genetic contributions to smoking, potential applications of this research for cessation treatment, and legal, ethical and social implications of future use of genotyping for cessation. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of OTC transdermal nicotine replacement therapy.
  Other Names: GES
  Arms: Genetic Education Session (GES)
Behavioral: Nutrition Education Session — To control for an attention placebo effect, the control group will receive information about nutritional guidelines as established by the USDA and the FDA. The attention control group will be referred to as the Nutritional Education Session (NES) group. The content of NES sessions one and two are use of the USDA (MyPyramid) dietary and food safety guidelines. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of OTC transdermal nicotine replacement therapy.
  Other Names: NES
  Arms: Nutrition Education Session (NES)

SUMMARY:
This study will test the effects of an educational program about genetics and smoking on smokers' thoughts, feelings, and behaviors before and after participating in smoking cessation treatment. This includes describing participants' knowledge about genetics and smoking, their use of strategies to stop smoking, and experiences when quitting smoking. This study will determine how smokers respond to information about genetics and smoking in anticipation of using genetic information to individualize pharmacological therapy for smoking cessation.

Two groups will participate in this study. The experimental group will participate in two educational sessions about genetics and smoking. The control group will participate in two educational sessions about nutrition. Both the experimental and control groups will participate in a standard, group smoking cessation program with 6 weeks of over-the-counter (OTC) transdermal nicotine replacement therapy. Assignment to either of the two groups is random.

The primary specific aim is to compare the effects of the experimental group to the attention control group on smoking-related mental representations, appraisals, behaviors, and affective responses over time. The secondary aim is to explore whether personality characteristics (trait negative affectivity and curiosity) and educational level moderate the effects of the genetic educational program on smoking-related mental representations, appraisals, behaviors, and affective responses. The hypotheses of the study are as follows:

1. When compared to the attention control group, the experimental group will demonstrate:

   * Smoking-Related Mental Representations:
   * Greater knowledge of genetic contributions to smoking
   * Greater endorsement of genetic contributions to smoking
   * More positive attitudes towards NRT
   * Increased abstainer and decreased smoker self-schemas
   * Smoking-Related Appraisal: greater perceived risk for genetic predispositions to smoking
   * Smoking-Related Behaviors: greater interest in genotyping.
2. When compared to the attention control group, the experimental group will differ in:

   * Smoking-Related Appraisals: self-efficacy for cessation and abstinence
   * Smoking-Related Behaviors: number of quit attempts, abstinence, nicotine dependence
   * Affective Responses: negative affect and intrusive/avoidant thoughts

DETAILED DESCRIPTION:
Background. Reducing cigarette smoking among adults is a major public health objective. Although the target prevalence for adult smoking is < 12% by 2010 (DHHS 2000), current estimates indicate that 20.8%, or 45.3 million adults, currently smoke (CDC, 2007). An estimated 44.2% of smokers tried to quit at least one day in the last 12 months (CDC, 2007), yet <10% of smokers who try to quit remain abstinent (Benowitz, 2008). Even with intensive treatment, only 11-20% of smokers are abstinent for 6 months (Sutherland, 2003). Smoking also results in an enormous economic burden, with health-care and lost productivity costs totaling approximately $167 billion per year (CDC, 2008). A limitation of current treatment guidelines is a lack of specificity for individual smokers. Completion of the sequencing of the human genome and the current focus on genomics (Collins, Green, Guttmacher, & Guyer, 2003) provides an unprecedented opportunity to study the biobehavioral factors influencing smoking. This research will contribute to individualized treatment by providing a better understanding of the effects of genetic, psychological, and environmental factors and their interaction on smoking initiation, maintenance, cessation, and relapse (Lerman, Schnoll & Munafo, 2007; Morgan et al., 2003; Swan et al., 2003). Both candidate gene studies to identify specific genes that affect smoking and pharmacogenomic studies that investigate the effects of selected genes on treatment response contribute to a growing body of knowledge about genetic influences on smoking. The anticipated outcome of these studies will be the ability to individualize type, dose, and duration of treatment based on smokers' genotypes (Lerman, Schnoll & Munafo). Ultimately, the long-term goal of this research is to decrease relapse and promote sustained abstinence.

The Genetic Education and Smoking Model provides a framework for investigating variables that potentially influence the ways smokers respond to information about: (a) genetic contributions to smoking and (b) the potential for genetically-informed cessation treatment. Based on social-cognitive theory and the Common Sense Model (CSM)(Cervone, 2004; Brownlee, Leventhal, & Leventhal, 2000), the Genetic Education and Smoking Model proposes that genetic education will influence smokers' mental representations and appraisals about genetics and smoking in addition to their smoking-related behaviors and affective responses.

As genetically-informed cessation treatment becomes a part of research and clinical care, smokers will need a degree of genetic literacy to make informed decisions (McInerney, 2002; Shields, Lerman, & Sullivan, 2004). There is a growing body of scientific knowledge to guide an educational program about genetic contributions to smoking and the potential for genetically-informed cessation treatment. Epidemiologic twin studies consistently support a genetic cause for smoking, with an estimated 56% of the variance for smoking initiation and 67% of progression to nicotine dependence due to additive genetic effects (Sullivan and Kendler, 1999). Findings from several genome-wide scans using linkage analysis have identified chromosomes 1, 2, 4, 5, 6, 9, 10, 11, 14, 17, 18, and 21 as containing possible susceptibility loci for smoking-related genes (Li,Cheng, Ma, & Swan, 2003; Li, Ma, & Beuten, 2004). Several candidate-genes for smoking heritability have been identified, including nicotinic acetylcholine receptors (nAChRs), dopamine receptor (DRD2 and DRD4) and transporter (SLC6A3) genes, the catechol-o-methyl-transferase (COMT) gene, the mu opioid receptor (OPRM1) gene, and the serotonin transporter (5-HTT) gene (Lerman, Schnoll, & Munafo, 2007; Schnoll, Johnson, & Lerman, 2007). Polymorphisms of CYP2A6, a cytochrome P450 enzyme, play a major role in the inactivation of nicotine to its metabolite, cotinine (Messina, Tyndale, & Sellers, 1997; Benowitz, 2008).

Specific Aims. The primary specific aim is to compare the effects of the experimental group to the attention control group on smoking-related mental representations, appraisals, behaviors, and affective responses over time. The primary aim will be achieved using a randomized, longitudinal, two-group repeated measures design to determine the direct effects of the intervention on smoking-related mental representations, appraisals, behaviors, and affective responses.

The secondary aim is to explore whether personality characteristics (trait negative affectivity and curiosity) and educational level moderate the effects of the genetic educational program on smoking-related mental representations, appraisals, behaviors, and affective responses.

The secondary aim will be achieved with multiple and logistic regression to determine whether personality traits and educational level moderate the effects of the intervention on the identified smoking-related outcomes.

Methods. Participants will be assigned randomly to either the experimental or attention control groups. The groups will be balanced for gender and number of cigarettes smoked per day using stratified randomization (Friedman, Furberg, & DeMets, 1996). Age and baseline data for major study variables will be treated as covariates.

The experimental group, referred to as the Genetic Education Session (GES) group, will receive education about two smoking-related genotypes, DRD2 and CYP2A6. The content of GES session one is basic genetics and includes concepts and terminology, the impact of the Human Genome Project on health-care and the use of genetic counseling and testing. The content of GES session two is research about smoking and genetics. The content focuses on the multifactorial nature of smoking; research findings about genetic contributions to smoking, specifically for candidate genotypes DRD2 and CYP2A6; and potential applications of this research for cessation treatment, including legal, ethical and social implications of genotyping. To control for an attention placebo effect (Meltzoff, 1998), the control group will receive information about nutritional guidelines as established by the U.S. Department of Agriculture (USDA) and FDA. The attention control group will be referred to as the Nutritional Education Session (NES) group. The content of NES sessions one and two are aimed at understanding and using dietary and food safety guidelines. Following the genetic or nutritional education sessions, both groups will receive a standard cognitive-behavioral smoking cessation intervention with NRT in the form of transdermal nicotine (TN) patch. This intervention will be referred to as the standard smoking cessation (SSC) sessions. SSC content focuses on the: (a) nature of nicotine addiction; (b) use of self-change strategies in the form of self-monitoring, stimulus identification and control, stress management, and relapse prevention; and (3) use of nicotine replacement to manage craving and withdrawal symptoms. The SSC sessions consists of four 2-hour group counseling sessions and one follow-up telephone call after the last session. The intervention will occur over a 5-week period after the GES or NES. Participants will receive a 6-week supply of TN patches in the following dosages: 21 mg/24hours for 4 weeks and 14 mg/24 hours for 2 weeks (Fiore Jaen, Baker al., 2008). A 1-week supply of patches will be distributed during SSC sessions 2-3 and a 2-week supply will be distributed at session 4. The final two weeks of free TN in 14 mg/24hours strength will be mailed to participants' homes during week 7. Participants will be encouraged to purchase a two-week supply of the 7 mg/24hours patches for the final two weeks of an 8-week course of TN. They will also have the option of using combination therapy as recommended in the 2008 guideline, to augment the TN with other NRT (gum, spray, inhaler) or bupropion SR. This option will be explained at the time of obtaining informed consent so participants can visit their primary care provider to obtain prescription medication (nicotine spray or inhaler or bupropion SR) prior to the SSC. Data will be collected on use of TN alone or in the recommended combinations. Expired air CO measurements will be conducted at each Session as feedback/motivation for participants. Session 1 CO measurement will be used as the baseline CO data.

Data Collection. Data collection in the form of self report questionnaires will occur at four time points, Time 1 through Time 4 (T1-T4). Baseline data collection (T1) will be followed by randomization to the experimental or control group. T2 data will be collected in two parts (T2a&b) to obtain initial post-intervention data for variables pertaining to each of these sessions: T2a will occur at the end of the education sessions (GES or NES) and T2b will occur at the end of the SSC sessions (i.e., 6 weeks). T2a Questionnaires will be distributed at the end of these sessions and return by the start of the SSC (Week 3). T2b questionnaires will be distributed at the end of the SSC. Questionnaires will be returned by postage-paid mail by Week 8. If needed, participants will be reminded to do this at the follow-up telephone session. Two additional data collections (T3-T4) will occur at twelve weeks and 6 months after the end of the SSC. T3-T4 data will consist of self-report questionnaires and in-person measurement of expired air CO with salivary cotinine verification of abstinence for participants not using NRT and whose CO measurement is <8-10 ppm (Benowitz et al., 2002).

Data Analysis. Preliminary analyses of the dependent variables will include frequency distributions to look for outliers, descriptive statistics and plots to assess normality, and bivariate scatterplots to evaluate linearity of relationships among study variables. Statistical methods of dealing with nonnormality, such as transformations of the raw data, may be employed prior to analysis. For all scales, internal consistency reliability coefficients will be estimated. All primary analyses will be based on an intent-to-treat paradigm. Each participant's data will be analyzed according to their randomized assignment, regardless of whether they completed all intervention sessions. The analysis plan will be carried out in order to work out any methodological issues, but because this is not a fully powered study, significant findings are not expected at the .05 level. A more liberal level of .10 will be used for significance tests, and emphasis will be placed on descriptive statistics and estimating effect sizes.

For Aim 1, the primary endpoint of mean change over time relative to baseline will be compared for the experimental and control groups using Generalized Estimating Equations (GEE) methodology (Laing & Zeger, 1986). A model will be fit incorporating terms to test the effects of the intervention and time, covarying for baseline values, for age, and for amount smoked. An interaction term will also be included to test whether the rate of change over time is the same for both groups. If difficulties occur with implementing GEE because of the relatively small number of cohorts per group in the pilot study, the model may be simplified to a cross-sectional analysis with individuals nested within cohorts at each time point.

For Aim 2, multiple and logistic regression will be used to predict the outcome variables from the independent variables and tests of moderation will be conducted according to procedures described by Baron & Kenny (1986).

ELIGIBILITY:
Inclusion Criteria:

* Current Smoker
* Smoking ten or more cigarettes per day
* 19 years or older
* Intention of quitting smoking in the next month
* Agree to use two forms of acceptable birth control while using the nicotine replacement patch

Exclusion Criteria:

* Not currently seeking treatment for a mental disorder with psychotic symptoms
* Not currently pregnant nor nursing
* Not been recently diagnosed or currently affected with cancer or any other life-threatening illness
* No recent heart attack
* No history of high blood pressure or not currently receiving treatment to manage high blood pressure
* No history of an irregular heartbeat
* Not currently taking medications to help quit smoking (i.e. Chantix, Zyban or Wellbutrin, NRT)
* No history of adverse effects from using nicotine replacement patches
* Not currently experiencing serious pain or discomfort due to heart disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-02-01; Primary Completion 2012-04-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia F Houfek, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to all researchers in both the private and public sector free or for a nominal charge with minimal restrictions via computerized data file from the research team. A codebook identifying the dataset variables will also be made available. The final dataset will not contain protected health information (PHI). Researchers requesting data must agree to the conditions of use governing access to the public release of data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution to third parties, and proper acknowledgement of the data resource. The data will be made available no later than acceptance for publication of the main findings from the final dataset.
Supporting Information: Analytic Code
Time Frame: After main study findings are published.
Access Criteria: Researchers in the public or private sector studying genetic education for smoking cessation who contact the PI.

REFERENCES:
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Benowitz NL. Clinical pharmacology of nicotine: implications for understanding, preventing, and treating tobacco addiction. Clin Pharmacol Ther. 2008 Apr;83(4):531-41. doi: 10.1038/clpt.2008.3. Epub 2008 Feb 27. PMID 18305452
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Cervone D. The architecture of personality. Psychol Rev. 2004 Jan;111(1):183-204. doi: 10.1037/0033-295X.111.1.183. PMID 14756593
- [Background] Collins FS, Green ED, Guttmacher AE, Guyer MS; US National Human Genome Research Institute. A vision for the future of genomics research. Nature. 2003 Apr 24;422(6934):835-47. doi: 10.1038/nature01626. Epub 2003 Apr 14. No abstract available. PMID 12695777
- [Background] Stewart SL, Cardinez CJ, Richardson LC, Norman L, Kaufmann R, Pechacek TF, Thompson TD, Weir HK, Sabatino SA; Centers for Disease Control and Prevention (CDC). Surveillance for cancers associated with tobacco use--United States, 1999-2004. MMWR Surveill Summ. 2008 Sep 5;57(8):1-33. PMID 18772853
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2006. MMWR Morb Mortal Wkly Rep. 2007 Nov 9;56(44):1157-61. PMID 17989644
- [Background] Brownlee, S., Leventhal, H., & Leventhal, E. A. (2000). Regulation, self-regulation, and construction of the self in maintenance of physical health. In M. Boekaerts, P.R. Pintrich, & M. Zeidner, (Eds.). Handbook of Self-Regulation. San Diego, CA: Academic Press, pp. 369-416.
- [Background] Department of Health & Human Services (DHHS). (2000). Healthy People 2010: Understanding and improving health. Conference edition. Washington, DC: U.S. Government Printing Office.
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] Friedman, L.M., Furberg, C.D., & DeMets, D.L. (1996). Fundamentals of Clinical Trials. 3rd ed. St.Louis: Mosby.
- [Background] Lerman CE, Schnoll RA, Munafo MR. Genetics and smoking cessation improving outcomes in smokers at risk. Am J Prev Med. 2007 Dec;33(6 Suppl):S398-405. doi: 10.1016/j.amepre.2007.09.006. PMID 18021915
- [Background] Li MD, Ma JZ, Beuten J. Progress in searching for susceptibility loci and genes for smoking-related behaviour. Clin Genet. 2004 Nov;66(5):382-92. doi: 10.1111/j.1399-0004.2004.00302.x. PMID 15479180
- [Background] Li MD, Cheng R, Ma JZ, Swan GE. A meta-analysis of estimated genetic and environmental effects on smoking behavior in male and female adult twins. Addiction. 2003 Jan;98(1):23-31. doi: 10.1046/j.1360-0443.2003.00295.x. PMID 12492752
- [Background] Liang, K.Y., & Zeger, S.L. (1986). Longitudinal data analysis using generalized linear models. Biometrika, 73, 13-22.
- [Background] Swan GE, Hudmon KS, Jack LM, Hemberger K, Carmelli D, Khroyan TV, Ring HZ, Hops H, Andrews JA, Tildesley E, McBride D, Benowitz N, Webster C, Wilhelmsen KC, Feiler HS, Koenig B, Caron L, Illes J, Cheng LS. Environmental and genetic determinants of tobacco use: methodology for a multidisciplinary, longitudinal family-based investigation. Cancer Epidemiol Biomarkers Prev. 2003 Oct;12(10):994-1005. PMID 14578134
- [Background] Sutherland, B.A. (2003). Evidence for counseling effectiveness for smoking cessation. Journal of Clinical Psychiatry Monograph, 18, 22-34.
- [Background] Sullivan PF, Kendler KS. The genetic epidemiology of smoking. Nicotine Tob Res. 1999;1 Suppl 2:S51-7; discussion S69-70. doi: 10.1080/14622299050011811. PMID 11768187
- [Background] Shields A, Lerman C, Sullivan P. Translating emerging research on the genetics of smoking into clinical practice: ethical and social considerations. Nicotine Tob Res. 2004 Aug;6(4):675-88. doi: 10.1080/14622200410001734058. PMID 15370164
- [Background] McInerney J. Education in a genomic world. J Med Philos. 2002 Jun;27(3):369-90. doi: 10.1076/jmep.27.3.369.2977. PMID 12187440
- [Background] Meltzoff, J. (1998). Critical Thinking about Research. Washington, DC: American Psychological Association.
- [Background] Messina ES, Tyndale RF, Sellers EM. A major role for CYP2A6 in nicotine C-oxidation by human liver microsomes. J Pharmacol Exp Ther. 1997 Sep;282(3):1608-14. PMID 9316878
- [Background] Morgan GD, Kobus K, Gerlach KK, Neighbors C, Lerman C, Abrams DB, Rimer BK. Facilitating transdisciplinary research: the experience of the transdisciplinary tobacco use research centers. Nicotine Tob Res. 2003 Dec;5 Suppl 1:S11-9. doi: 10.1080/14622200310001625537. PMID 14668084
- [Background] Schnoll RA, Johnson TA, Lerman C. Genetics and smoking behavior. Curr Psychiatry Rep. 2007 Oct;9(5):349-57. doi: 10.1007/s11920-007-0045-3. PMID 17915073

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We had 103 participants in the study. The last 14 participants were recruited at the end of the funding period and had a shortened intervention and data collection protocol to determine feasibility of the shortened protocol. The main study variables were analyzed on 89 participants (50 in the experimental GES group; 39 in the attentional control NES group) who completed the original protocol.
Groups:
- Genetic Education Session (GES): The objectives are to: discuss the impact of the human genome project; define basic genetic concepts and terminology; distinguish between single-gene and multifactorial genetic diseases/conditions; describe genetic counseling/testing; identify uses of pharmacogenetics; discuss psychological and legal/ethical implications of genetic discoveries; smoking as a multifactorial behavior; findings of epidemiological studies about smoking heritability; research about candidate genotypes dopamine D2 receptor (DRD2) and CYP2A6; and potential use of genotyping to tailor smoking cessation treatment.
  Genetic Education Session: The intervention includes receiving education about genetics and smoking. The content is basic genetics and education about the multifactorial nature of smoking; research findings about genetic contributions to smoking, potential applications of this research for cessation treatment, and legal, ethical and social implications of future use of genotyping for cessation. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of over-the-counter (OTC) transdermal nicotine replacement therapy.
- Nutrition Education Session (NES): Nutrition Education Session: To control for an attention placebo effect, the control group will receive information about nutritional guidelines as established by the USDA and the FDA. The attention control group will be referred to as the Nutritional Education Session (NES) group. The content of NES sessions one and two are use of the U.S. Department of Agriculture (USDA) (MyPyramid) dietary and food safety guidelines. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of over-the-counter (OTC) transdermal nicotine replacement therapy.
Period: Overall Study
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES)
Started | 57 | 46
Started Original Protocol (This milestone indicates the number of participants included in the original protocol.) | 50 | 39
Completed Original Protocol (This milestone indicates the number of participants who completed the original protocol.) | 10 | 12
Completed (This row indicates the number of participants who completed the study (i.e., both the original protocol and the revised protocol that occurred at the end of the funding period) as stated in the Pre-Assignment Details.) | 11 (11 participants in the experimental (GES) arm completed the study, of which 10 completed the original protocol.) | 17 (17 participants in the control group (NES) completed the study, of which 12 completed the original protocol.)
Not Completed | 46 | 29
Not completed — Withdrawal by Subject | 46 | 29

BASELINE CHARACTERISTICS:
Groups:
- Genetic Education Session (GES): The objectives are to: discuss the impact of the human genome project; define basic genetic concepts and terminology; distinguish between single-gene and multifactorial genetic diseases/conditions; describe genetic counseling/testing; identify uses of pharmacogenetics; discuss psychological and legal/ethical implications of genetic discoveries; smoking as a multifactorial behavior; findings of epidemiological studies about smoking heritability; research about candidate genotypes DRD2 and CYP2A6; and potential use of genotyping to tailor smoking cessation treatment.
  Genetic Education Session: The intervention includes receiving education about genetics and smoking. The content is basic genetics and education about the multifactorial nature of smoking; research findings about genetic contributions to smoking, potential applications of this research for cessation treatment, and legal, ethical and social implications of future use of genotyping for cessation. All participants also receive a 5-week standard cognitive-behavioral smoking cessation intervention with 6 weeks of OTC transdermal nicotine replacement therapy.
- Total: Total of all reporting groups
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES) | Total
Number analyzed (Participants) | 57 | 46 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 46 | 100
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 31 | 17 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 51 | 42 | 93
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 46 | 103

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Genetic Contributions to Smoking
Description: Knowledge of genetic contributions to smoking. Name of Scale: Genetic Knowledge Test (9 items). Minimum/Maximum Scores: 0-9. Higher score means better outcome.
Time Frame: One week after completion of the two Educational Sessions (GES or NES). Educational sessions occurred over two weeks.
Population: Analysis is based on the number of participants who completed the two educational sessions, i.e., GES for the experimental group and NES for the attentional control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES)
Number analyzed (Participants) | 44 | 33
score on a scale
  Baseline | 5.25 (2.55) | 3.73 (2.66)
  End of Educational Sessions | 7.04 (1.72) | 4.03 (2.78)
Statistical Analysis 1: Comparison: Genetic Education Session (GES) vs Nutrition Education Session (NES); The scores on the Genetic Knowledge Test for both groups between baseline and the end of the educational sessions were analyzed with repeated measures ANOVA; Test type: Other; p < 0.01, ANOVA — A priori threshold for the P-Value was.05 or less

2. Primary Outcome: Smoking-Related Appraisals
Description: Self-efficacy for Quitting/Resisting Smoking. Self-efficacy/Temptation Scale (Velicer, DiClemente, Rossi & Prochaska, 1990) Total Score. Scores range from 1 to 5, with higher scores indicating greater self-efficacy. Source: Velicer, W.F., DiClemente, C.C., Rossi, J.S., & Prochaska, J.O. (1990). Relapse situations and self-efficacy: An integrative model. Addictive Behaviors, 15, 271-283.
Time Frame: Six weeks after the baseline data collection, which was the end of the Smoking Cession Sessions.
Population: Analysis is based on the number of participants who completed the Smoking Cessation Sessions and returned questionnaire data for the following time points: baseline, end of the Educational Sessions, and end of the Smoking Cessation Sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES)
Number analyzed (Participants) | 28 | 24
score on a scale
  Baseline | 3.93 (.46) | 3.99 (.70)
  End of Educational Sessions | 3.80 (.60) | 3.86 (.69)
  End of Smoking Cessation Sessions | 2.73 (.86) | 2.57 (1.03)
Statistical Analysis 1: Comparison: Genetic Education Session (GES) vs Nutrition Education Session (NES); Data for Self-Efficacy for Quitting/Resisting Smoking were analyzed with repeated measures ANOVA using three time points: baseline, end of the educational sessions, and end of the smoking cessation sessions; Test type: Other; p = 0.44, ANOVA — The a priori threshold for statistical significance was a P-Value of .05 or less

3. Primary Outcome: Smoking Abstinence at End of Smoking Cessation Sessions
Description: Number of participants reporting Smoking Abstinence at the end of the Smoking Cessation Sessions and who had a carbon monoxide (CO) measurement of 6 ppm or less.
Time Frame: Six weeks, which was the end of the Smoking Cessation Sessions.
Population: Analysis based on the number of participants who completed the Smoking Cessation Sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES)
Number analyzed (Participants) | 28 | 25
Participants
  Number of Participants Quit | 11 | 10
  Number of Participants Not Quit | 17 | 15
Statistical Analysis 1: Comparison: Genetic Education Session (GES) vs Nutrition Education Session (NES); Test type: Other — Nominal data were analyzed with Chi Square; p = .88, Chi-squared — The a priori threshold P-Value for statistical significance was .05 or less

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Arm/Group | Genetic Education Session (GES) | Nutrition Education Session (NES)
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/46
Other Adverse Events (participants affected / at risk) | 0/57 | 0/46

LIMITATIONS AND CAVEATS:
Group sessions may have hindered attendance/study withdrawal. Of the 89 participants only 44 Experimental and 34 Control group participants received the GES or NES and 33 Experimental and 28 Control group participants completed the smoking cessation program. Future studies can determine if one session of GES/NES and individual smoking cessation sessions increases participation/retention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No